CLINICAL TRIAL: NCT05174741
Title: Effects of Pulmonary Rehabilitation Therapy on Pulmonary Function and Health Related Quality of Life in Non-chronic Obstructive Pulmonary Disease Patients
Brief Title: Pulmonary Rehabilitation in Non-chronic Obstructive Pulmonary Disease Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/00882 Aleena Ashraf
Record Dates: First submitted 2021-06-21; First posted 2022-01-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Pulmonary Fibrosis; Tuberculosis; Bronchiectasis; Asthma
Keywords: non-COPD; quality of life; pulmonary function
MeSH Terms: conditions — Pneumonia; Pulmonary Fibrosis; Tuberculosis; Bronchiectasis; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Chest Physiotherapy (Active Comparator): Diaphragmatic Breathing exercise 15 repetition ACBT *3 sets/session*TD Walk (10-15 minutes) * BD
  Interventions: Other: Conventional Chest Physiotherapy
- Aerobic Training group (Experimental): Supervised Conventional chest physiotherapy+ Aerobic training Conventional chest physiotherapy supervised (1st week) Then non supervised for 2nd to 6th week Warm-up (5 minutes) Breathing exercise and stepping Diaphragmatic Breathing exercise *15 Reps* TD
  Aerobic training on cycle ergometer:
  between 50% and 70% Vo2max, perceived exertion up to 11 on Borg scale 20-30 min/session/day Cool down (5 minutes) AROM +Body stretch
  Interventions: Other: Aerobic training Group

INTERVENTIONS:
Other: Conventional Chest Physiotherapy — Diaphragmatic Breathing exercise 15 repetition ACBT *3 sets/session*TD Walk (10-15 minutes) * BD
  Arms: Conventional Chest Physiotherapy
Other: Aerobic training Group — Supervised Conventional Chest Physiotherapy + Aerobic training
  Aerobic training on cycle ergometer:
  between 50% and 70% Vo2max, perceived exertion up to 11 on Borg scale 20-30 min/session/day
  Arms: Aerobic Training group

SUMMARY:
To determine the effect of pulmonary rehabilitation on pulmonary function in non-chronic obstructive pulmonary disease patients.To determine the effect of pulmonary rehabilitation on health related quality of life in non-chronic obstructive pulmonary disease patients.Limited researches are available in non chronic obstructive pulmonary disease patients.

DETAILED DESCRIPTION:
A review state that "Interstitial lung disease presents clinical features of exertional desaturation and a nonproductive cough. Patients with ILD have significantly reduced exercise capacity as manifested by a reduced maximum work load achieved during exercise, as well as a reduced maximal oxygen uptake VO2max." in previous studies Pulmonary rehabilitation is the use of exercise, education and behavioral interventions for diseases such as non-ILD restrictive lung disease, asthma, lung cancer, bronchiectasis , and pulmonary hypertension, pre and post op thoracic surgery patients.

Quality of life (QOL) as an individual's perception of contentment or satisfaction with life in areas he or she considers important, and we define health-related quality of life (HRQL) as an individual's perception of the impact of health (in all its many facets) on his or her quality of life. a study on pulmonary rehabilitation outcomes between individuals with chronic obstructive lung disease (COPD) and non-COPD disease and its impact on gender.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of non-COPD disease interstitial lung disease (pulmonary fibrosis), restrictive lung disease (TB, pneumonia), Bronchiectasis, and Asthma with FEV1 below 50%, FVC<80%, and FEV1/FVC>70%

Exclusion Criteria:

* Clinically/vitally unstable or having Uncontrolled DM/HTN, Current smokers or ex-smokers of less than 1 year.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 3 weeks, 6 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 3 weeks,6 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 3 weeks,6 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

SECONDARY OUTCOMES:
Health related Quality of life | 3 weeks,6 weeks
  Measured through St. George's Respiratory Questionnaire in its COPD-specific version (SGRQ-C). The SGRQ-C with 40 items provides three component scores for symptoms, activity and impact, and a total score. Each score ranges from 0 (no impairment) to 100 (worst possible). A difference of 4 unit points is considered the minimum clinically important difference (MCID).

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Pakistan railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No